CLINICAL TRIAL: NCT07201727
Title: Early Clinical Study of CD123+CLL-1 Dual-target CAR-T Cells Sequential Infusion CD7 CAR-T Cells and Bridging to Allogeneic Hematopoietic Stem Cell Transplantation for the Treatment of Relapsed and Refractory Acute Myeloid Leukemia
Brief Title: CD123+CLL-1 CAR-T Sequential Infusion With CD7 CAR-T and Bridging to Allo-HSCT for Relapsed/Refractory Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025079
Record Dates: First submitted 2025-09-05; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: AML - Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; CAR-T; Allogeneic hematopoietic stem cell transplantation; CD7; CD123; CLL1; CD123+CLL1
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD123+CLL-1 CAR-T sequential infusion with CD7 CAR-T and bridging to allo-HSCT (Experimental): Treat with CD123+CLL-1 dual-target CAR-T (JY017), then sequentially infuse CD7-targeted CAR-T (JY008) for patients not achieving MRD negativity, perform allo-HSCT based on patient conditions.
  Interventions: Biological: CD123+CLL-1 dual-target CAR-T cells sequential infusion CD7 CAR-T cells and bridging to allogeneic

INTERVENTIONS:
Biological: CD123+CLL-1 dual-target CAR-T cells sequential infusion CD7 CAR-T cells and bridging to allogeneic — For patients with refractory and relapsed AML, CD123+CLL-1 dual-target CAR-T cells (JY017) are used for treatment. Then, for patients who cannot achieve the minimum residual negative, CD7-targeted CAR-T cells (JY008) are sequentially infused. Finally, allogeneic hematopoietic stem cell transplantation is performed based on patient conditions.

SUMMARY:
This study is a single-arm, open-label, prospective clinical trial, with patients suffering from refractory and relapsed acute myeloid leukemia as the subjects. It plans to enroll 10 cases to evaluate the safety and efficacy of sequential CD123+CLL-1 CAR-T cells followed by CD7 CAR-T cells treatment.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, prospective clinical trial. It targets patients with relapsed/refractory acute myeloid leukemia (AML), planning to enroll 10 cases. The study will follow up and observe data related to adverse reactions and treatment efficacy after medication, aiming to evaluate the safety and efficacy of sequential therapy with two types of CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria：

* Patients are clinically diagnosed with relapsed or refractory acute myeloid leukemia；
* Tumor cells are confirmed to be CD123 or CLL-1 positive by flow cytometry (FCM) or immunohistochemistry, with a positivity rate of no less than 80%；
* Patients aged 18 to 75 years (inclusive)；
* The expected survival time is more than 3 months from the date of signing the informed consent;
* KPS≥80 points;
* The functions of vital organs need to meet the following conditions: ①LVEF>50%，and electrocardiogram is normal; ② Oxygen saturation ≥90%;③ SCr≤2.5ULN；④ALT and AST≤5ULN，TBil≤3ULN；
* Subjects intending to conceive must agree to use contraception prior to study enrollment and for six months post-study. In the event of pregnancy or suspected pregnancy, they should promptly notify the investigator.
* The subject or guardian understands and signs the Informed Consent Form (ICF).

Exclusion Criteria:

Any of the following conditions will not be eligible for enrolment in this study:

* Within one - year prior to signing the informed consent form, there is a history of heart failure of New York Heart Association (NYHA) class ≥ III, or myocardial infarction, cardiac angioplasty or stent implantation, unstable angina pectoris, or other cardiac diseases with prominent clinical symptoms, or the QTc interval is > 480 ms during screening (the QTc interval is calculated by the Fridericia formula);
* Those with active GvHD or those who need to use immunosuppressants;
* Patients who have had any malignancy other than acute myeloid leukemia (AML) within the past 5 years, except for those with adequately treated cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin, locally resected prostate cancer, or resected ductal carcinoma in situ of the breast;
* Patients who have active infections requiring systemic treatment or uncontrollable infections within 7 days prior to screening, except for mild urinary and genital infections and upper respiratory infections;
* There has been a history of autoimmune diseases (such as rheumatoid arthritis, systemic lupus erythematosus, Crohn's disease) that require systemic immunosuppressive/systemic disease regulatory drugs for treatment within the past two years;
* When screening, if the hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HbcAb) is positive and the peripheral blood hepatitis B virus (HBV) DNA is higher than the detection limit, it needs to be excluded. If the hepatitis C virus (HCV) antibody is positive, those with positive HCV RNA in peripheral blood need to be excluded. Those who are positive for human immunodeficiency virus (HIV) antibodies; Those who test positive for cytomegalovirus (CMV) DNA; Those with positive DNA test for lymphotropic human herpesvirus (EBV); Those who test positive for Treponema pallidum specific antibody (TPPA) need to be excluded;
* Participation in another clinical trial within 4 weeks or within 5 half-lives of the last dose of the drug from the previous clinical trial (whichever is longer);
* Has a history of severe allergy to biological products;
* Unstable systemic diseases as judged by the investigator: including but not limited to severe liver, kidney or metabolic diseases requiring medical treatment;
* Pregnant or lactating women, female subjects who plan to become pregnant within 2 years after CAR-T cell infusion, or male subjects whose partners plan to become pregnant within 2 years after their CAR-T cell infusion;
* conditions that the investigator believes may increase the risk to the subject or interfere with the results of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Monitor and record adverse events | From CAR - T cell infusion to 2 years later.

SECONDARY OUTCOMES:
Overall Response Rate | From CAR - T cell infusion to 2 years later .